CLINICAL TRIAL: NCT03520296
Title: Descriptive Study on the Evaluation of Well-being in Relation to Diet and Nutrition and Comparison Between Three Care Units in the Dijon University Hospital Centre
Acronym: ALIMS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BRINDISI UB 2016
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-04

CONDITIONS: Hospitalization in Cardiology, Orthopaedic Surgery or Endocrinology Departments
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients hospitalized in the cardiology unit
  Interventions: Other: Questionnaire
- Patients hospitalized in the orthopedic surgery unit
  Interventions: Other: Questionnaire
- Patients hospitalized in the endocrinology unit
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire evaluating well-being in relation to diet and nutrition

SUMMARY:
The aim of this study is to qualify patient well-being in relation to diet. The notion of dietary well-being is believed to be subjective and we wish to base it on tangible parameters (presentation of meals, variety of menus, social interaction, environment, convenience, pleasure...) in order to establish a score of dietary well-being that we will then correlate to the patient's nutritional status. This tool can then be used more widely as an assessment tool within health institutions.

ELIGIBILITY:
Inclusion Criteria:

* person who has given oral consent
* adult
* persons admitted to cardiology, orthopaedic surgery and endocrinology units
* absence of cognitive problems
* oral food intake

Exclusion Criteria:

* no affiliation to a national health insurance scheme
* current pregnancy
* blended diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in cardiology, orthopaedic surgery or endocrinology departments
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Questionnaire evaluating well-being in relation to diet and nutrition | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France